CLINICAL TRIAL: NCT00226655
Title: An Open-Labeled, Extended-Use of Human Corticotropin-Releasing Factor (hCRF) Intended for Patients Who Participate in Dexamethasone-Sparing Studies NTI 0302, NTI 0303, or Other Designated Studies
Brief Title: An Open-Labeled, Extended-Use of XERECEPT (hCRF) for Patients in Studies NTI 0302, 0303, or Other Designated Studies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celtic Pharma Development Services (Industry)
Collaborators: Neurobiological Technologies (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTI 0501
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Results first posted 2012-08-31 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-07

CONDITIONS: Brain Edema; Brain Tumor
Keywords: peritumoral brain edema; edema; malignant brain tumor; astrocytoma; brain tumor; dexamethasone; Decadron
MeSH Terms: conditions — Brain Edema; Brain Neoplasms; Edema; Astrocytoma | interventions — Corticotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- I (Experimental): All patients will receive hCRF (XERECEPT) 2mg/day
  Interventions: Drug: hCRF [XERECEPT (corticorelin acetate injection)]

INTERVENTIONS:
Drug: hCRF [XERECEPT (corticorelin acetate injection)] — 2mg/day
  Other Names: hCRF, XERECEPT (corticorelin acetate injection)

SUMMARY:
The purpose of this study is to examine the long-term safety and tolerability of human corticotropin-releasing factor (hCRF), XERECEPT®, in patients requiring dexamethasone (Decadron) to treat peritumoral brain edema. This open-label, extended-use study is open to all patients who participate in either of the blinded studies, NTI 0302, NTI 0303, or other designated studies, including patients who may have discontinued blinded study medication early but completed the protocol-stipulated follow-up periods.

DETAILED DESCRIPTION:
XERECEPT® is not a potential treatment for cancer, but may reduce the edema associated with tumors and as a result, decrease neurological symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Participation in and completion of stipulated final follow-up periods for study NTI 0302, NTI 0303, or other designated studies.
* Have a Karnofsky Performance of > 50 at Baseline
* Capable of self-administration of subcutaneous injections twice daily or availability of assistance from caregiver.
* Ability to provide written informed consent or, if unable to provide, have a legal guardian or representative provide written informed consent.
* For women of childbearing potential: a negative serum pregnancy test at Baseline

Exclusion Criteria:

* Concurrent enrollment in any investigational drug or device study, other than NTI 0302, NTI 0303, or other designated studies.
* Systemic steroid use for any indication other than peritumoral brain edema.
* Use or intended use of dexamethasone as an anti-emetic during study.
* Clinical signs and symptoms of cerebral herniation.
* Serious concomitant cardiovascular, pulmonary, renal, gastrointestinal or endocrine metabolic disease which could put the patient at unusual risk during study participation.
* Confounding previous or concurrent neurological disorders that would interfere with adequate clinical evaluation.
* Clinically significant head injury or chronic seizure disorder, if the condition results in functional impairment or is likely to interfere with evaluations.(Maintenance anticonvulsant therapy is allowed)
* Central nervous system (CNS) infection.
* Pregnancy, breastfeeding and/or refusal to practice birth control while in study, for women of childbearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2005-07; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Shapiro, MD, Principal Investigator — Barrow Neurological Institute
Locations (32):
- United States (25):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Stanford University Medical Center, Palo Alto, California
  - UC Davis Medical Center, Division of Medical Oncology, Sacramento, California
  - UC San Diego Cancer Center, San Diego, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Colorado Neurological Institute Center for Brain & Spinal Tumors, Englewood, Colorado
  - Mayo Clinic, Jacksonville, Florida
  - Cancer Institute of Orlando, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Feinberg School of Medicine, Northwestern University, Chicago, Illinois
  - Evanston Northwestern Healthcare, Evanston, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Hermelin Brain Tumor Center, Henry Ford Hospital, Detroit, Michigan
  - Dent Neurologic Institute, Amherst, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - University Hematology Oncology Care, LLC, Cincinnati, Ohio
  - Good Samaritan Hospital, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - Oregon Clinic, Portland, Oregon
  - Virginia Mason Clinic, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (7):
  - Cross Cancer Institute, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - The Moncton Hospital, Moncton, New Brunswick
  - Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia
  - Caner Centre of Southwestern Ontario/ Kingston General Hospital, Kingston, Ontario
  - Ottawa Regional Cancer Center, Ottawa, Ontario
  - Sunnybrook and Women's College Health Sciences Center, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started February 2005;
Pre-assignment Details: Patients rolled-over from previous placebo controlled studies; open label study so no group assignment
Groups:
- hCRF: All patients will receive hCRF (XERECEPT) 2mg/day
Period: Overall Study
Arm/Group | hCRF
Started | 112
Completed | 33
Not Completed | 79
Not completed — Death | 13
Not completed — Withdrawal by Subject | 15
Not completed — Adverse Event | 35
Not completed — Physician Decision | 6
Not completed — Clinical deterioration | 10

BASELINE CHARACTERISTICS:
Arm/Group | hCRF
Number analyzed (Participants) | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 101
  >=65 years | 11
Age Continuous [Mean (Standard Deviation); unit: years] | 51.4 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 44
Region of Enrollment [Number; unit: participants]
  United States | 101
  Canada | 6
  Australia | 4
  New Zealand | 1

OUTCOME MEASURES:

1. Primary Outcome: Long Term Safety and Tolerability of hCRF
Description: Number of patients reporting adverse events
Time Frame: Prospective
Population: Intent to Treat
Measure: Number; unit: Participants
Groups:
- hCRF: hCRF administered 1mg bid subcutaneously
Arm/Group | hCRF
Number analyzed (Participants) | 112
Participants | 111 (4.5)

ADVERSE EVENTS:
Arm/Group | hCRF
Serious Adverse Events (participants affected / at risk) | 72/112
Other Adverse Events (participants affected / at risk) | 111/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | hCRF (N=112)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Blindness (Eye disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Injection site urticaria (General disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 4 (4)
Clostridial infection (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Perianal abscess (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5)
Rectal abscess (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 3 (3)
Septic shock (Infections and infestations) | 2 (2)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 4 (4)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5)
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myelodysplastic syndrom (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 25 (25)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1)
Brain stem haemorrhage (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Cerebrospinal fistula (Nervous system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 17 (17)
Encephalopathy (Nervous system disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 3 (3)
Status epilepticus (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Agitation (Psychiatric disorders) | 8 (8)
Confusional state (Psychiatric disorders) | 1 (1)
Mental state changes (Psychiatric disorders) | 2 (2)
Personality change (Psychiatric disorders) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 2 (2)
Rena tubular necrosis (Renal and urinary disorders) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | hCRF (N=112)
Diarrhoea (Gastrointestinal disorders) | 13 (13)
Nausea (Gastrointestinal disorders) | 23 (23)
Injection site erythema (General disorders) | 18 (18)
Oedema peripheral (General disorders) | 13 (13)
Cushingoid (Endocrine disorders) | 8 (8)
Vision blurred (Eye disorders) | 7 (7)
Constipation (Gastrointestinal disorders) | 11 (11)
Vomiting (Gastrointestinal disorders) | 12 (12)
Asthenia (General disorders) | 7 (7)
Fatigue (General disorders) | 23 (23)
Gait disturbance (General disorders) | 8 (8)
Pneumonia (Infections and infestations) | 9 (9)
Upper respiratory tract infection (Infections and infestations) | 9 (9)
Urinary tract infection (Infections and infestations) | 8 (8)
Contusion (Injury, poisoning and procedural complications) | 7 (7)
Alanine aminotransferase increased (Investigations) | 6 (6)
Weight decreased (Investigations) | 6 (6)
Anorexia (Metabolism and nutrition disorders) | 6 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 8 (8)
Fall (Injury, poisoning and procedural complications) | 12 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 14 (14)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7)
glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 34 (34)
Aphasia (Nervous system disorders) | 9 (9)
Convulsion (Nervous system disorders) | 32 (32)
Dizziness (Nervous system disorders) | 8 (8)
Headache (Nervous system disorders) | 30 (30)
Hemiparesis (Nervous system disorders) | 15 (15)
Hypoaesthesia (Nervous system disorders) | 10 (10)
Tremor (Nervous system disorders) | 7 (7)
Confusional state (Psychiatric disorders) | 11 (11)
Depression (Psychiatric disorders) | 6 (6)
Insomnia (Psychiatric disorders) | 11 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Rash (Skin and subcutaneous tissue disorders) | 8 (8)
Skin fragility (Skin and subcutaneous tissue disorders) | 7 (7)
Flushing (Vascular disorders) | 27 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less